CLINICAL TRIAL: NCT05556967
Title: Identification of Surrogate Blood and/or Urine Biomarker for Immulina TM in Normal Humans
Brief Title: Identification of Surrogate Blood and/or Urine Biomarker for Immulina TM (Trademark) in Normal Humans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-363; 1U19AT010838-01 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Adherence, Patient
Keywords: Immulina TM; Healthy Participants; Natural Dietary Supplement
MeSH Terms: conditions — Patient Compliance | interventions — Immulina

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immulina Dietary Supplementation (Experimental): Immulina Dietary Supplementation (200 mg per capsule) 4-200 mg capsules given by mouth once on the only study visit day.
  Interventions: Drug: Immulina

INTERVENTIONS:
Drug: Immulina — Immulina is a highly standardized extract derived from various preparations of Spirulina, a cyanobacterium, marketed as a dietary supplement and has been utilized in several clinical studies describing its immunopotentiating properties.
  Other Names: Spirulina

SUMMARY:
This is a pilot study for identifying plasma and/or urine-derived adherence/surrogate biomarker candidates for verifying Immulina™ ingestion by human volunteers (collected before and after consumption of Immulina™, a natural dietary supplement).

DETAILED DESCRIPTION:
This pilot study is interventional, and all participants will receive one 800 mg dose of Immulina™ (four 200 mg capsules), a natural supplement, after a baseline blood and urine collection, then follow with 1 hour, 3 hour and 6 hour post-Immulina™ blood and urine collections. Samples will be sent to UM National Center for Natural Products Research (NCNPR) to analyze and compare timed blood and urine samples using gas chromatography and liquid chromatography to detect volatile and non-volatile compounds, gamma-linolenic acid (GLA), sulfoquinovose (SQ), 5'-methylsulfinyladenosine (MSA), palmitic acid, linoleic acid, palmitoleic acid and oleic acid to screen the chemical fingerprints of the human samples. The mean of the 7 biomarkers for the 4 time points will be measured and compared.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18-50 years old
* If female of childbearing potential, using acceptable means of birth control or postmenopausal for at least two years
* Healthy

Exclusion Criteria:

* pregnant or lactating females
* significant acute disease
* recurrent medications for chronic disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
gamma-linolenic acid (GLA), ug/mL | Over 7 hour period
  Differences in GLA between baseline, 1 hour post-Immulina, 3 hour post-Immulina and 6 hour post-Immulina
Sulfoquinovose (SQ), ug/mL | Over 7 hour period
  Differences in SQ between baseline, 1 hour post-Immulina, 3 hour post-Immulina and 6 hour post-Immulina
5'-methylsulfinyladenosine (MSA), ug/mL | Over 7 hour period
  Differences in MSA between baseline, 1 hour post-Immulina, 3 hour post-Immulina and 6 hour post-Immulina
palmitic acid, ug/mL | Over 7 hour period
  Differences in palmitic acid between baseline, 1 hour post-Immulina, 3 hour post-Immulina and 6 hour post-Immulina
linoleic acid, ug/mL | Over 7 hour period
  Differences in linoleic acid between baseline, 1 hour post-Immulina, 3 hour post-Immulina and 6 hour post-Immulina
palmitoleic acid, ug/mL | Over 7 hour period
  Differences in palmitoleic acid between baseline, 1 hour post-Immulina, 3 hour post-Immulina and 6 hour post-Immulina
steric acid, ug/mL | Over 7 hour period
  Differences in steric acid between baseline, 1 hour post-Immulina, 3 hour post-Immulina and 6 hour post-Immulina
oleic acid, ug/mL | Over 7 hour period
  Differences in oleic acid between baseline, 1 hour post-Immulina, 3 hour post-Immulina and 6 hour post-Immulina

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, Jr., MD, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Clinical Research and Trials Unit - University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu D, Meydani M, Leka LS, Nightingale Z, Handelman GJ, Blumberg JB, Meydani SN. Effect of dietary supplementation with black currant seed oil on the immune response of healthy elderly subjects. Am J Clin Nutr. 1999 Oct;70(4):536-43. doi: 10.1093/ajcn/70.4.536. PMID 10500023
- [Background] Tahvonen RL, Schwab US, Linderborg KM, Mykkanen HM, Kallio HP. Black currant seed oil and fish oil supplements differ in their effects on fatty acid profiles of plasma lipids, and concentrations of serum total and lipoprotein lipids, plasma glucose and insulin. J Nutr Biochem. 2005 Jun;16(6):353-9. doi: 10.1016/j.jnutbio.2005.01.004. PMID 15936647
- [Background] Geppert J, Demmelmair H, Hornstra G, Koletzko B. Co-supplementation of healthy women with fish oil and evening primrose oil increases plasma docosahexaenoic acid, gamma-linolenic acid and dihomo-gamma-linolenic acid levels without reducing arachidonic acid concentrations. Br J Nutr. 2008 Feb;99(2):360-9. doi: 10.1017/S0007114507801577. Epub 2007 Aug 3. PMID 17678567
- [Background] Martens-Lobenhoffer J, Meyer FP. Pharmacokinetic data of gamma-linolenic acid in healthy volunteers after the administration of evening primrose oil (Epogam). Int J Clin Pharmacol Ther. 1998 Jul;36(7):363-6. PMID 9707349
- [Background] Xue, C.; Hu, Y.; Saito, H.; Zhang, Z.; Li, Z.; Cai, Y.; Ou, C.; Lin, H.; Imbs, A. B. Molecular species composition of glycolipids from Sprirulina platensis. Food Chemistry 2002, 77 (1), 9-13.
- [Background] Goddard-Borger ED, Williams SJ. Sulfoquinovose in the biosphere: occurrence, metabolism and functions. Biochem J. 2017 Feb 20;474(5):827-849. doi: 10.1042/BCJ20160508. PMID 28219973
- [Background] Mills, J. S.; Mills, G. C.; Mcadoo, D. J. Isolation and identification of 5'-methylthioadenosine sulfoxide from human urine. Nucleosides and Nucleotides 1983, 2 (5), 465-478.